CLINICAL TRIAL: NCT05703672
Title: 4th Generation E-cigarettes: Reducing Harm and Quitting Combustible Cigarettes in Dual Users
Brief Title: Switching to E-cigarettes in Smokers Not Interested in Quitting
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STUDY00146887
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Smoking Reduction
MeSH Terms: conditions — Smoking Reduction | interventions — Varenicline; Electronic Nicotine Delivery Systems

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Varenicline and electronic cigarette (Experimental): At the end of the 6-week open label phase, dual users of cigarettes and e-cigarettes will receive 1mg varenicline to take twice daily for 12 weeks. They will also receive an additional 12 weeks of the nicotine salt-based pod system e-cigarette.
  Interventions: Drug: Varenicline Tartrate; Other: Electronic cigarette
- Placebo and electronic cigarette (Placebo Comparator): At the end of the 6-week open label phase, dual users of cigarettes and e-cigarettes will receive placebo pills to take twice daily for 12 weeks. They will also receive an additional 12 weeks of the nicotine salt-based pod system e-cigarette.
  Interventions: Drug: Placebo; Other: Electronic cigarette
- Open label electronic cigarette (Other): All participants will receive an initial 6-week supply of the study electronic cigarette.
  Interventions: Other: Electronic cigarette

INTERVENTIONS:
Drug: Varenicline Tartrate — 0.5 mg once daily for days 1-3, 0.5mg twice daily for days 4-7 and 1.0 mg twice daily from day 8 through week 12.
  Arms: Varenicline and electronic cigarette
Drug: Placebo — One pill (white) once daily for days 1-3, one pill (white) twice daily for days 4-7 and one pill (blue) twice daily from day 8 through week 12.
  Arms: Placebo and electronic cigarette
Other: Electronic cigarette — Nicotine salt pod based e-cigarette in 5% nicotine

SUMMARY:
The objectives of this application are to 1) compare short- and long-term harm reduction and abuse liability potential of a nicotine salt pod-based electronic cigarettes (EC) in adult (AA) exclusive EC, dual cig-EC, and exclusive cig users, 2) characterize factors that predict who switches fully, partially, or not at all, and 3) examine if harm reduction can be further enhanced by treating dual users with varenicline (VAR) to eliminate cigarette smoking.

DETAILED DESCRIPTION:
Adult cigarette smokers (n=500) who are interested in switching to a nicotine salt-based electronic cigarette (EC) and are not established EC users will receive a 6-week supply of the EC and assistance with switching. After six weeks, those that are dual users (n=221) will receive an additional 12 weeks of the EC and be randomized in a 2:1 fashion to receive 12 weeks of varenicline (VAR) or placebo (PBO) and additional counseling to support a complete switch. Follow-up for all participants will continue through week 52. The primary outcome is change in the potent lung carcinogen, NNAL, between exclusive EC, dual cig-EC, and exclusive cig users at week 6.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 21 years of age
* Smoke >5 cigarettes per day
* Smoked cigarettes for > 6 months
* Verified smoker (CO > 5 ppm)
* Functioning telephone
* Interested in switching to EC
* Willing to take varenicline and complete all study visits

Exclusion Criteria:

* Interested in quitting smoking
* Use of smoking cessation pharmacotherapy in the month prior to enrollment
* Use of other tobacco products in past 30 days (i.e., cigarillos, cigars, hookah, smokeless tobacco, pipes)
* EC use on > 4 of the past 30 days
* Uncontrolled hypertension: BP > 180 (systolic) or > 105 (diastolic)
* Heart-related event in the past 30 days
* Medical contraindications to VAR: unstable cardiac condition (e.g., unstable angina or AMI) cardiac event, or stroke in the past 4 weeks; renal impairment; history of clinically significant allergic reactions; history of epilepsy or seizure disorder; hospitalized for psychiatric issue in past 30 days; active suicidal ideation
* Pregnant, contemplating getting pregnant, or breastfeeding
* Plans to move from Kansas City metro area during the treatment and follow-up phase
* Another household member enrolled in the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2026-12-07 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Reduction in toxicant exposure as measured by NNAL (4- (methylnitrosamino)-1-(3-pyridyl)-1-butanol) . | Week 6
  Reduction in toxicant exposure as measured by NNAL excretion from baseline to week 6.

SECONDARY OUTCOMES:
Carbon Monoxide (CO) verified 7-day point prevalence abstinence from cigarettes | Week 12 post randomization
  CO verified 7-day point prevalence abstinence from cigarettes at week 12 post randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Nollen, PhD, Principal Investigator — University of Kanas Medical Center
Locations (2):
- United States (2):
  - Swope Health Central, Kansas City, Missouri
  - University of Kansas Medical Center, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: No